CLINICAL TRIAL: NCT04023942
Title: Lifestyle Intervention Study
Brief Title: Personalized Nutrition and EHealth: Lifestyle Intervention (LION) Study for Weight Loss Maintenance
Acronym: LION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Christina Holzapfel, Principal investigator, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01EA1709
Record Dates: First submitted 2019-07-11; First posted 2019-07-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Weight maintenance; Lifestyle intervention; Dietary intervention; Formula diet; App; Newsletter; Digital tool; Low carb; Low fat; Meal challenges
MeSH Terms: conditions — Obesity; Weight Loss; Alzheimer Disease | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: This clinical study is a single-center 2*2 factorial randomized trial. For the weight maintenance step, participants will be randomized into one of the four weight maintenance intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low carb - App-based group (Active Comparator): Low carb is defined as 30 energy percent from carbs and consist of 20 energy percent from protein. The daily energy requirement is calculated for each participant individually, based on his/hers resting metabolic rate and physical activity level. Daily energy intake should be 10% lower than the calculated daily energy requirement. Participants assigned to the app-based group works together with a personal coach via app, providing nutritional guidance and support during the 12-month weight maintenance step.
  Interventions: Behavioral: Weight maintenance intervention
- Low carb - Newsletter-based group (Active Comparator): Low carb is defined as 30 energy percent from carbs and consist of 20 energy percent from protein. The daily energy requirement is calculated for each participant individually, based on his/hers resting metabolic rate and physical activity level. Daily energy intake should be 10% lower than the calculated daily energy requirement. The newsletter intervention group gets regularly digital newsletters, in the same frequency as "contacts" take place in the app-based group.
  Interventions: Behavioral: Weight maintenance intervention
- Low fat - App-based group (Active Comparator): Low fat is defined as 25 energy percent from fat and consist of 20 energy percent from protein. The daily energy requirement is calculated for each participant individually, based on his/hers resting metabolic rate and physical activity level. Daily energy intake should be 10% lower than the calculated daily energy requirement. Participants assigned to the app-based group works together with a personal coach via app, providing nutritional guidance and support during the 12-month weight maintenance step.
  Interventions: Behavioral: Weight maintenance intervention
- Low fat - Newsletter-based group (Active Comparator): Low fat is defined as 25 energy percent from fat and consist of 20 energy percent from protein. The daily energy requirement is calculated for each participant individually, based on his/hers resting metabolic rate and physical activity level. Daily energy intake should be 10% lower than the calculated daily energy requirement. The newsletter intervention group gets regularly digital newsletters, in the same frequency as "contacts" take place in the app-based group.
  Interventions: Behavioral: Weight maintenance intervention

INTERVENTIONS:
Behavioral: Weight maintenance intervention — Weight maintenance intervention (52 weeks): After randomization, participants will follow either a low carb or a low fat diet and get nutritional assistance either by an app or a newsletter, based on the group they got randomized to (low carb/app, low carb/newsletter, low fat/app, low fat/newsletter).
  Other Names: Dietary Intervention

SUMMARY:
Despite standardized intervention strategies, weight loss and weight loss maintenance largely differ from person to person. Factors which may contribute to these individual differences is current object of research.

In order to investigate predictors and barriers for weight management and to investigate two different dietary interventions and two different digital tools for weight maintenance, the LION-Study was designed as follows: Step I (screening, baseline phenotyping), step II (weight loss intervention with formula diet), step III (weight maintenance intervention with 4 intervention groups: low carb/newsletter; low carb/app; low fat/newsletter; low fat/app) and step IV (follow-up). Participants are required to attend visits at seven time points.

At screening (month 0) a telephone-based screening interview takes place, in order to test eligibility of the potential participant. If the person is eligible, two consecutive baseline face-to-face visits are planned during step I. After completion of the eight weeks weight loss intervention (month 3), an additional visit takes place followed by three consecutive visits in the weight maintenance step (month 6, 9 and 15). The study ends with a final visit after the follow-up (month 27). Additional contacts (face-to-face and telephone) take place during the weight loss intervention step. Participants will regularly receive a bag with the required formula diet meals. During these "pick up" appointments, the study team actively get in face-to-face contact with participants.

At the different visits, data are collected by questionnaires, medical investigations (e.g. MRI, motor function, resting metabolic rate), blood withdrawal as well as urine, feces and saliva sampling.

Primary objective is to evaluate the effect of two diets (low carb/low fat) and two digital tools (app/newsletter) on long-term weight loss maintenance 12 months after weight loss.

Secondary objective is to identify genetic, epigenetic, physiological, psychological and lifestyle factors that predict the success of weight loss and weight loss maintenance.

DETAILED DESCRIPTION:
Step I - Screening and baseline phenotyping When a potential suitable participant is interested, a screening interview to check eligibility will take place by phone after oral agreement is given. The structured screening interview is carried out by means of a questionnaire in the format of a Case Report Form (CRF). Suitable persons are provided with participant´s information and data protection sheet and with the "declaration of consent". Sufficient time for consideration is given between the screening interview and visit 1A, where written consent is signed.

After the telephone-based screening interview, eligible participants are required to provide written consent. Participants will undergo clinical examinations at two visits (V1A + V1B), serving primarily for phenotyping as well as for detection of potentially unknown exclusion criteria. The order of some measurements carried out during V1A and V1B as well as the type of lipid challenge is randomized.

Data collection V1A:

* Resting metabolic rate
* Metabolic response to meal challenge
* Anthropometry
* Vital parameters
* Blood parameters
* Clinical, lifestyle (nutrition, physical activity), psychological, environmental and social factors (questionnaires and protocols)
* Sampling of blood samples for further research questions

Data collection V1B:

* Metabolic response to meal challenge
* Vital parameters
* Blood parameters
* Urine parameters
* Hand Strength Measurement
* Clinical, lifestyle (nutrition, physical activity), psychological, environmental and social factors (questionnaires and protocols)
* Sampling of blood, urine and saliva
* Optional: Adipose tissue distribution by MRI measurement; parameters for physical strength, motor function and body static condition; 24h urine collection; fecal samples

Step II - Weight loss intervention Once participant is still deemed eligible after V1A and V1B, the formula-based low calorie diet (LCD) starts as weight loss intervention. Formula products will be provided once per week. An additional daily intake of 200 g raw or cooked non-starchy vegetables is allowed. Participants fulfill a food diary to record eaten products including drinks and vegetables and to record well-being or side effects. Furthermore, participants are phenotyped by a continuous glucose measurement during the first four weeks of intervention.

Data collection V2:

* Anthropometry
* Vital parameters
* Blood and urine parameters
* Clinical, lifestyle (nutrition, physical activity), psychological, environmental and social factors (questionnaires and protocols)
* Resting metabolic rate
* Hand strength measurement
* Documentation of safety
* Continuous glucose measurement
* Sampling of blood, urine, and saliva
* Optional: Adipose tissue distribution by MRI measurement; parameters for physical strength, motor function and body static condition; 24h urine collection; fecal samples Step III - Weight maintenance intervention

If weight loss is > 4 kg after eight weeks, the participant is eligible for randomization into one of the following four weight maintenance intervention arms:

Low carb - App-based group Low carb - Newsletter-based group Low fat - App-based group Low fat - Newsletter-based group

Data collection V3A:

* Anthropometry
* Blood and urine parameters
* Clinical, lifestyle (nutrition, physical activity), psychological, environmental and social factors (questionnaires and protocols)
* Documentation of safety
* Sampling of blood and urine samples for further research questions, e.g. metabolic profile (to be confirmed)
* Optional: 24h urine collection

Data collection V3B:

* Anthropometry
* Blood parameters
* Clinical, lifestyle (nutrition, physical activity), psychological, environmental and social factors (questionnaires and protocols)
* Documentation of safety
* Sampling of blood samples for further research questions, e.g. metabolic profile (to be confirmed)

Data collection V3C:

* Anthropometry
* Blood and urine parameters
* Resting metabolic rate
* Vital parameters
* Clinical, lifestyle (nutrition, physical activity), psychological, environmental and social factors (questionnaires and protocols)
* Documentation of safety
* Hand strength measurement
* Sampling of blood, urine, and saliva
* Optional: Adipose tissue distribution by MRI measurement; parameters for physical strength, motor function and body static condition; 24h urine collection; fecal samples Step IV - Follow-up During follow-up, all participants receive the same newsletters with nutritional information every 3 months (independent of weight maintenance intervention group). Further weight management is carried out by "self-help".

Data collection V4:

* Anthropometry
* Vital parameters
* Blood parameters (
* Clinical, lifestyle (nutrition, physical activity), psychological, environmental and social factors (questionnaires and protocols)
* Resting metabolic rate
* Sampling of blood

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years
* BMI: 30,0 - 39,9 kg/m2
* Owner of a smartphone
* Caucasian
* No severe diseases
* Informed written consent

Exclusion Criteria:

* Diabetes mellitus
* Severe cardiovascular and/or respiratory disease
* Untreated high blood pressure
* Severe kidney disease
* Active cancer (or in remission)
* Inflammatory bowel disease
* Severe chronic infections and/or inflammations
* Severe mental-health disorders
* Neurodegenerative disorders
* Endocrine diseases
* Lipedema
* Pregnancy and lactation
* Vigorous weight fluctuations (> 5 kg) in the last 3 months
* Immobility
* Surgery in the last 3 months
* Participation in other intervention studies
* Carrier of pace makers
* Blood donation or transfusion in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Weight maintenance 12 months after weight loss intervention | 15 months
  Body weight change in kg and % (from baseline weight)

SECONDARY OUTCOMES:
Weight change after eight weeks of formula diet | month 3
  Body weight in kg and % (from baseline weight)
Glucose | month 0, 3, 6, 9, 12, 15, 27
  Change in glucose in mg/dl
Insulin | month 0, 3, 6, 9, 12, 15, 27
  Change in insulin in µU/ml
Lipids | month 0, 3, 6, 9, 12, 15, 27
  Change in blood lipids (total cholesterin, triglyzeride, HDL cholesterin, LDL cholesterin - highly correlated to each other) in mg/dl
Leptin | month 0, 3, 6, 9, 12, 15, 27
  Change in leptin in ng/ml
Resting metabolic rate | month 0, 3, 15, 27
  Resting metabolic rate in kilocalories / 24 hours
Magnetic resonance imaging (MRI) | month 0, 3, 15, 27
  MRI data (organ volume, proton density fat fraction)
Insulin response on meal challenges | month 0
  Insulin response at different time points during meal challenge in µU/ml
Glucose response on meal challenges | month 0
  Glucose response at different time points during meal challenge in mg/dl
Lipid response on meal challenges | month 0
  Lipid (total cholesterin, triglyzeride, HDL cholesterin, LDL cholesterin - highly correlated to each other) response at different time points during meal challenge in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Christina Holzapfel, PhD, Principal Investigator — TUM School of Medicine, Technical University of Munich
Locations (1):
- Institute for Nutritional Medicine, Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
We will apply principles which meet standards of findability, accessibility, interoperability, and reusability (FAIR) in the management of data in our project. The owner of the data will be the Institute for Nutritional Medicine at TUM School of Medicine, Technical University of Munich. The data and samples will be safely stored for long term and can be easily accessed and/or downloaded by the study team. For collaboration partners defined dataset and samples will be provided with well-defined license and access conditions.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: On request participant data collected during the trial, after deidentification and according to informed consent. Researches who provide a methodologically sound proposal. On request to principle investigator (Christina Holzapfel, christina.holzapfel@tum.de).

REFERENCES:
- [Background] Reik A, Schauberger G, Wiechert M, Hauner H, Holzapfel C. Association Between the Postprandial Response to an Oral Glucose Tolerance Test and Anthropometric Changes After an 8-Week Low-Calorie Formula Diet - Results From the Lifestyle Intervention (LION) Study. Mol Nutr Food Res. 2024 Jun;68(12):e2400106. doi: 10.1002/mnfr.202400106. Epub 2024 Jun 8. PMID 38850172
- [Background] Reik A, Holzapfel C. Randomized Controlled Lifestyle Intervention (LION) Study for Weight Loss and Maintenance in Adults With Obesity-Design and Methods. Front Nutr. 2020 Nov 10;7:586985. doi: 10.3389/fnut.2020.586985. eCollection 2020. PMID 33240920
- [Background] Junker D, Wu M, Reik A, Raspe J, Rupp S, Han J, Nabauer SM, Wiechert M, Somasundaram A, Burian E, Waschulzik B, Makowski MR, Hauner H, Holzapfel C, Karampinos DC. Impact of baseline adipose tissue characteristics on change in adipose tissue volume during a low calorie diet in people with obesity-results from the LION study. Int J Obes (Lond). 2024 Sep;48(9):1332-1341. doi: 10.1038/s41366-024-01568-6. Epub 2024 Jun 26. PMID 38926461
- [Background] Somasundaram A, Wu M, Reik A, Rupp S, Han J, Naebauer S, Junker D, Patzelt L, Wiechert M, Zhao Y, Rueckert D, Hauner H, Holzapfel C, Karampinos DC. Evaluating Sex-specific Differences in Abdominal Fat Volume and Proton Density Fat Fraction at MRI Using Automated nnU-Net-based Segmentation. Radiol Artif Intell. 2024 Jul;6(4):e230471. doi: 10.1148/ryai.230471. PMID 38809148